CLINICAL TRIAL: NCT06730503
Title: Sugar Chain Heterogeneity in Immunotherapy Response and Efficacy Prediction of Lung Cancer
Brief Title: Glycoprotein in Immunotherapy Response and Efficacy Prediction of Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xiaomin Niu, Principal Investigator, Shanghai Chest Hospital
Other Study IDs: THORACIC006
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; immunotherapy; Immune checkpoint inhibitors; PD-L1; resistance; sugar chain heterogeneity; glycoprotein
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The blood specimens are stored in the refrigerator at -20°C or -80°C as specified in the clinical trial protocol. Test specimens and backup specimens should be kept in separate refrigerators to prevent malfunction of one of the refrigerators. Centrifugation time, specimen collection and specimen storage time should be carried out in strict accordance with the requirements of the clinical trial protocol.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anti-PD-1/PD-L1 monoclonal antibody
  Interventions: Drug: Immune checkpoint inhibitor

INTERVENTIONS:
Drug: Immune checkpoint inhibitor — Observe a situation before and after immunotherapy

SUMMARY:
Immunotherapy has improved the prognosis of non-small cell lung cancer (NSCLC) patients, but about 80% of patients do not respond at all (primary resistance), and some patients initially respond to immunotherapy, later relapse and develop disease progression (acquired resistance).

So the objective of this research is to explore the sugar chain heterogeneity of primary and acquired resistance to immunotherapy in patients with NSCLC.

DETAILED DESCRIPTION:
Immunotherapy has improved the prognosis of non-small cell lung cancer (NSCLC) patients, but about 80% of patients do not respond at all, which is called primary resistance. Absence of the PD-L1 expression is regarded as one of primary resistant reasons to immunotherapy, there are some other reasons which have been reported to be related with the primary resistance, including tumor mutation burden (TMB), microsatellite instability (MSI), tumor neoantigen burden (TNB), HLA genotype, loss of heterozygosity (LOH), intra tumoral heterogeneity (ITH), genome wide doubling (WGD), and ploidy. While some patients initially respond to immunotherapy, later relapse and develop disease progression, which is called acquired resistance, like escaping of interferon signaling pathways or mutations in some important genes such as B2M/JAK1/JAK2.

Sugar chains, as the third chain of life except nucleic acids and proteins. More than half of the proteins in the human body have sugar chain modifications. During the occurrence, development, and metastasis of malignant tumors such as lung cancer, colorectal cancer, and gastric cancer, protein glycosylation undergoes corresponding changes as the disease progresses. Discovering and elucidating disease-related glycoproteins and their characteristic sugar chains is of great significance for searching for disease-specific biomarkers.

So the objective of this research is to explore the comprehensive characteristic sugar chain markers of primary and acquired resistance to immunotherapy in patients with Chinese advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Be able to provide informed consent, and understand and agree to follow the research requirements;
* Advanced non-small cell lung cancer;
* Patients receiving immune checkpoint inhibitor treatment represented by anti-PD-1/PD-L1 monoclonal antibody;
* The patient must be able to provide 10mL peripheral whole blood samples before- and after- ICIs;
* ECOG physical fitness status ≤1;
* The patient must have at least one measurable lesion (assessed according to RECIST v1.1);
* Life expectancy ≥ 12 weeks;
* The patient must have adequate organ function, and must be reached absolute neutrophil count (ANC) ≥1.5x10^9/L, platelets ≥100x10^9/L, hemoglobin ≥90g/L, international normalized ratio (INR) or prothrombin time ≤ 1.5x ULN , activated partial thromboplastin time (aPTT)≤1.5x ULN, serum total bilirubin≤1.5x ULN (Patients with Gilbert syndrome can be enrolled if total bilirubin<3x ULN), Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤2.5x ULN(Patient with liver metastases, this standard is AST and ALT≤5x ULN) within 7 days before treatment;

Exclusion Criteria:

* Patients with other tumors. Except for basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin or cervical cancer in situ, subjects who have received potential radical treatment and have not relapsed within 5 years before the start of treatment can be included in the study;
* Have received any approved systemic anti-tumor immunotherapy before starting the research treatment;
* A history of interstitial lung disease, non-infectious pneumonia or uncontrolled systemic diseases, including diabetes, hypertension, pulmonary fibrosis, acute lung disease, etc.;
* Severe chronic or active infections that require systemic antibacterial, antifungal or antiviral therapy, including tuberculosis infection;
* Known human immunodeficiency virus infection; previous allogeneic stem cell transplantation or organ transplantation;
* The investigator judged that the patient's compliance during the study period was insufficient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients with advanced NSCLC patients receiving immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 5 years
  The investigator (and the chief radiologist) used the RECIST 1.1 evaluation criteria to evaluate the efficacy indicators. CT or MRI imaging data of the chest and abdomen collected regularly during the screening/baseline period and the study period were used for tumor evaluation. Only when there may be primary or metastatic disease in the pelvis, pelvic imaging is recommended. Any other disease-affected areas (for example, the pelvis and brain) should undergo additional imaging studies based on the individual patient's signs and symptoms. If an unplanned evaluation is performed and it is shown that the patient has not progressed, follow-up evaluation should be performed at the next scheduled visit as much as possible. Scanning/tumor evaluation continued throughout the study period until RECIST 1.1 appeared
Progression-free survival (PFS) | Up to 5 years
  Calculate the time from the immunotherapy to the tumor progression/all-cause death/the end of the follow-up period.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 5 years
  Calculate the time from the immunotherapy to the end of the all-cause death/follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaomin Niu, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided